CLINICAL TRIAL: NCT03602495
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study of Donafenib in Patients With Radioiodine-Refractory Differentiated Thyroid Cancer
Brief Title: A Phase 3 Study of Donafenib in Patients With Radioiodine-refractory Differentiated Thyroid Cancer
Acronym: DTC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on IDMC's recommendations during the interim analysis"the trial has reached the goal of early termination of the trial". the sponsor communicating with CDE, CDE agreed to unblind the trial and submit a NDA.
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZGDD3
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Differentiated Thyroid Cancer
MeSH Terms: interventions — donafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donafenib (Experimental): Participants randomly assigned in a 2:1 ratio to receive blinded study drug (Donafenib or matching placebo) until documentation of disease progression (confirmed by IRC), development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Donafenib
- Placebo (Placebo Comparator): Participants randomly assigned in a 2:1 ratio to receive blinded study drug (Donafenib or matching placebo) until documentation of disease progression (confirmed by IRC), development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donafenib — Donafenib 0.3g Bid orally, continuously. Dose interruptions or reductions were allowed for subjects who experienced treatment-related toxicity.
  Arms: Donafenib
Drug: Placebo — Matching placebo Bid orally, continuously.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 3 study to compare the progression free survival, overall response rate (ORR) and safety of participants treated with Donafenib 0.3g Bid by continuous oral dosing versus placebo.

DETAILED DESCRIPTION:
Blinded Phase: Participants will receive blinded study drug (Donafenib/placebo) in 2:1 ratio until documentation of disease progression (confirmed by independent imaging review committee), development of unacceptable toxicity, or withdrawal of consent. After having completed the primary analysis, subjects treated with Donafenib who have not experienced disease progression may request to continue open label Donafenib at the same dose, according to the clinical judgment of the investigator. Participants who discontinue treatment for any reason other than disease progression will be followed in the Blinded Phase until disease progression or start of another anticancer treatment; these participants then enter the Open label Phase for survival follow-up.

Open label Phase: Participants in the placebo arm who have disease progression confirmed by IRC could request to enter the Optional Open Label Donafenib Treatment Period and receive Donafenib treatment. Participants will receive Donafenib treatment until disease progression, development of intolerable toxicity, or withdrawal of consent. Participants who had disease progression during the blinded Phase and did not enter the Optional Open Label Donafenib Treatment Period and all participants who discontinued Donafenib treatment in the Optional Open Label Donafenib Treatment Period will enter the follow-up period. Participants will be followed for survival, and all anticancer treatments will be recorded until the time of death.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥18 years;
* Advanced or metastases thyroid cancer;
* Histologically or cytologically confirmed diagnosis of one of the following differentiated thyroid cancer (DTC) subtypes: papillary thyroid cancer, follicular thyroid cancer or Hurthle cell, poorly differentiated carcinoma;
* Disease progression within 14 months prior to randomization.
* Measurable disease according to (RECIST 1.1) and Have a minimum of one measurable lesion.
* Subjects must be 131I-refractory / resistant as defined by at least one of the following:

  1. One or more measurable lesions that do not demonstrate iodine uptake on any radio-iodine scan
  2. One or more measurable lesions that has progressed by RECIST 1.1 within 14 months of 131I therapy, despite demonstration of radio-iodine avidity at the time of that treatment by pre-treatment scanning.
  3. Cumulative activity of 131I of >600 mCi or 22 gigabequerels (GBq)
* Subjects may have not received molecular targeted therapy;
* Subjects with known brain metastases who have completed whole brain radiotherapy, stereotactic radiosurgery or complete surgical resection, will be eligible if they have remained clinically stable, asymptomatic and off of steroids for one month
* Subjects must tolerate to thyroxin ,and TSH suppression (TSH less than 0.5 mU/mL);
* Before 14 days prior to study entry,(before laboratory examination for 14days no blood transfusion,not use albumin and Hematopoietic Stimulating Factor),Adequate laboratory examination :

  1. Absolute neutrophil count (ANC) greater than or equal to 1500/ mm3;
  2. Platelets greater than or equal to 100,000/mm3 ;
  3. Hemoglobin greater than or equal to 9.0g/dL
  4. Adequate blood coagulation function:International Normalized Ratio(INR)≤2.
  5. Adequate liver function: Bilirubin less than or equal to 1.5 x the upper limit of normal(ULN) ;Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 2.5 x the upper limit of normal (ULN),for liver metastasis ALT and AST less than or equal to 5.0 x the upper limit of normal (ULN);
  6. serum creatinine less than or equal to 1.5 x the upper limit of normal (ULN);creatinine clearance less than 50ml/min
* Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0~2；
* Life expectancy ≥12 weeks;
* All females must have a negative serum or urine pregnancy test. Females of childbearing potential and male subjects who are partners of women of childbearing potential must use or their partners must use a highly effective method of contraception;
* Voluntary provision of written informed consent and the willingness and ability to comply with all aspects of the protocol.
* Swallow oral drugs and keep them in the body.

Exclusion Criteria:

* Other pathologic subtypes of the thyroid, Anaplastic or medullary carcinoma of the thyroid etc;
* Prior treatment to TKI or other molecular targeted drugs；
* Subjects who have received any chemotherapy or extra radiotherapy（in addition to low dose chemotherapy for radiosensitization） within 4 weeks prior to randomization and should have recovered from any toxicity related to previous anti-cancer treatment;
* Known or suspect to TKI food allergy;in the study be allergic to drugs;
* Active malignancy (except for differentiated thyroid carcinoma, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 5 years;
* Major surgery, open biopsy or severe trauma within 4 weeks prior to the first dose of study drug;
* An unhealed wound, ulcer, or fracture;
* Evidence of bleeding and coagulation disorders;
* Using the antiplatelet drugs(except for a small dose of aspirin which is not more than 100mg)；
* The risk of Infiltration and bleeding of the trachea, bronchi and esophagus，not using topical treatment berore randomize;
* Bleeding of more than Grade 3 within 3 months prior to the first dose of study drug;
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug;
* Cardiac arrhythmia requiring medical treatment,QTc more than 480ms；Adequately controlled blood pressure with or without antihypertensive medications, defined as BP less than 140/90 mmHg using at least 2 kinds of medicine;
* Venous or arterial thromboembolic events，cerebral blood-vessel accident，arterial thrombosis，pulmonary embolism，deep-venous thrombosis，within 6 months of the first dose of study drug;
* Active infection more than Grade 2 (any infection requiring treatment);
* All chemotherapy or radiation-related toxicities must have resolved to less than Grade 2 severity, except alopecia neurotoxicity;
* HIV infectious,active infection of the HCV and HBV (HBV-DNA more than 1000 copise/ml，expect the chronic asymptomatic HBV carrier);
* Epileptic seizure being drug treatment;
* Using the strong - acting CYP3A4 inducer(phenytoin,carbamazepine,rifampicin,rifapentine,phenobarbital) within 7 days of the first dose of study drug;
* using biological reaction regulator(g-csf granulocyte colony stimulating factor) within 21 days of the first dose of study drug;
* The drug abuse,medicine,psychology and social disease which may be have an effect on study result;
* Any malabsorption disease;
* The disease which is unstable and harm to safty and research compliance of patient;
* Take the other clinical research treatment in the study and within 4 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Date of randomization to the date of disease progression or death (whichever occurred first) or up to approximately 3 years.
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression or death (whichever occurred first), as determined by Independent imaging review committee(IRC) using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 for the double-blind treatment period.

SECONDARY OUTCOMES:
Overall Survival (OS) | Date of randomization until date of death from any cause, or up to approximately 3 years.
  Overall survival measured from the date of randomization until date of death from any cause.
Objective Response Rate(ORR) | From randomization of the first subject until the last subject complete 24 months treatment
  ORR is defined as the percentage of subjects with total number of Complete Response(CR)+total number of Partial Response(PR).
Disease Control Rate(DCR) | From randomization of the first subject until the last subject complete 24 months treatment
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Time To Disease Progression (TTP) | From randomization of the first subject until the last subject complete 24 months treatment
  TTP was defined as the time from date of randomization to disease progression radiological. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yan Song, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun D, Zhang X, Jin X, Shi C, Sun Y, Zhang Y, Liang J, Lin Y. BRAFV600E mutation is associated with better prognoses in radioactive iodine refractory thyroid cancer patients treated with multi-kinase inhibitors: a retrospective analysis of registered clinical trials. Thyroid Res. 2025 Feb 10;18(1):5. doi: 10.1186/s13044-025-00223-0. PMID 39924483